CLINICAL TRIAL: NCT05303701
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Design, Prospective, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Subcutaneous Administration of GV1001 1.12 mg/Day in Patients With Moderate to Severe Alzheimer Disease
Brief Title: GV1001 Subcutaneous for the Treatment of Moderate to Severe Alzheimer's Disease(AD)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GV1001-AD-CL3-S002
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Moderate to Severe Alzheimer's Disease
Keywords: Alzheimer's Disease; GV1001
MeSH Terms: conditions — Alzheimer Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GV1001 Placebo (Placebo Comparator): GV1001 placebo (0.9% saline) subcutaneous injection will be administered once a week for 4 weeks and then administered every 2 weeks for 20 weeks in a double-blind phase.
  During the open-label extension phase, patients assigned to the GV1001 Placebo arm in the double-blind phase will receive a placebo in the first week, followed by 1.12 mg of GV1001 weekly for 4 weeks and then every 2 weeks until EOT (End of Treatment).
  Interventions: Drug: GV1001 Placebo; Drug: GV1001 1.12mg
- GV1001 1.12 mg (Experimental): GV1001 1.12 mg subcutaneous injection will be administered once a week for 4 weeks and then administered every 2 weeks for 20 weeks in a double blind phase.
  During the open-label extension phase, patients will alternate between 1.12 mg of GV1001 and placebo weekly for the first 5 weeks to maintain double blindness, and then 1.12mg of GV1001 every 2 weeks until EOT.
  Interventions: Drug: GV1001 Placebo; Drug: GV1001 1.12mg

INTERVENTIONS:
Drug: GV1001 Placebo — 0.9% normal saline
  Other Names: Normal saline
Drug: GV1001 1.12mg — Lyophilized peptide from hTERT
  Other Names: Tertomotide 1.68mg

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of GV1001 administered subcutaneously in patients with moderate to severe Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Studies using in vivo and in vitro Alzheimer's Disease (AD) models have shown that GV1001 inhibits neurotoxicity, apoptosis, and the production of reactive oxygen species induced by amyloid beta (Aβ) in neural stem cells by mimicking the extra-telomeric functions of human telomerase reverse transcriptase (hTERT). In nonclinical studies, using both mild (early stage) and severe (late stage) AD mouse models, GV1001 was shown to improve cognitive function and memory, as well as significantly reduce the amount of Aβ and tau proteins. The multifunctional effect of GV1001 makes it a promising therapeutic option for the treatment for AD. In a completed Phase 2 study (NCT03184467) conducted in Korea, GV1001 showed significant improvement in change from baseline of Severe Impairment Battery score at Week 24 and demonstrated a clinically acceptable safety profile in patients with moderate to severe AD.

This is a multi-center, randomized, double-blinded, placebo-controlled, parallel design, prospective phase 3 study in participants with moderate to severe AD. The study consists of 24 weeks of Double-blind phase and 25 weeks of open-label phase.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 55 to ≤ 85 years
2. Subjects who satisfy diagnostic criteria for dementia in DSM-IV (Diagnostic and Statistical Manual of Mental Disorders Fourth edition)
3. Subjects who are clinically diagnosed with probable Alzheimer's disease as defined in the NINCDS-ADRDA (National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association) criteria
4. Subjects with a K-MMSE (Korea Mini-Mental State Examination) score ≤ 19 at the screening visit
5. Subjects with GDS (Global Deterioration Scale) grade 5 to 6
6. Subjects who have no other diseases to cause dementia other than AD as a result of MRI or CT scan within 12 months from the screening visit
7. Subjects who are taking donepezil alone or donepezil and memantine in combination at a stable dose without a dose change over 3 months before screening
8. Subjects who are not illiterate
9. Subjects who can walk with or without assist device to visit hospitals or clinics to undergo cognitive tests and other tests
10. Subjects with caregiver who can accompany all visits with the subjects as scheduled for this trial, supervise subject's compliance for the tests and examination process and provide information about the subject's indications, and who give written consent
11. Subjects and/or caregivers who voluntarily agreed in written to participate in the clinical trial

Exclusion Criteria:

1. Subjects who have other causes of dementia as listed below according to CT/MRI test and neurologic examination within 12 months of screening or at the time of screening.

   * Subjects with possible, probable or definite vascular dementia according to NINDS-AIREN (National Institute of Neurological Disorders and Stroke and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences) criteria
   * Subjects with other central nervous system diseases that can cause the impairment of cognitive function (cerebrovascular disease including cerebrovascular dementia, Parkinsonism, Huntington's disease, subdural hematoma, normal pressure hydrocephalus, brain tumor, Creutzfeldt-Jakob disease, etc.)
   * Subjects with neuropathy such as delusion, delirium, epilepsy, etc.
2. Subjects who have abnormal test results which are considered to contribute to the severity of their dementia or be the cause of dementia in the vitamin B12, folic acid, syphilis serology, and the thyroid stimulating hormone (TSH) tests
3. Subjects who have a history of significant psychiatric illness such as schizophrenia or bipolar affective disorders which may interfere with the participation of this clinical trial according to the investigator's judgment or who are suffering from depression
4. Subjects with a history of known or suspected seizures including febrile seizure, recent loss of consciousness which is not explained or history of significant head trauma accompanied by loss of consciousness
5. Subjects in any medical condition that may interfere with the evaluation and progression of the clinical trial according to the investigator's judgment (acute or unstable cardiovascular disease, uncontrolled hypertension (>160/100 mmHg) at Visit 1 and Visit 2, insulin-dependent or uncontrolled diabetes at Visit 1 (HbA1c> 8% on screening test), etc.).
6. Subjects who are hypersensitive to the components of the investigational product.
7. Subjects with a history of alcohol and drug abuse or dependence (except nicotine dependence) within the last 2 years.
8. Subjects with a history of cancer within the past 5 years (however, non-metastatic skin basal cell carcinoma and/or skin squamous cell carcinoma, carcinoma in suit of uterine cervix or non-progressive prostate cancer may be acceptable and If cancer is considered to have been treated at the judgement of the investigator, if subjects are not taking anticancer or radiation therapy and are considered that treatment is not required for the next 5 years at the discretion of the investigator, enrollment is possible)
9. Subjects with renal dysfunction (Creatinine Clearance (Clcr) < 30 mL/min)
10. Subjects with serious hepatic dysfunction (Alanine aminotransferase or Aspartate aminotransferase ≥ 2.0 normal upper limit)
11. Subjects who are taking prohibited drugs or expected to be administered during clinical trial period

    * Drugs for the treatment of Alzheimer's Disease or other cognitive impairment other than donepezil and memantine
    * Anticholinergic drugs (local usages are allowable, such as pilocarpine eye drops), antidepressant drugs (tricyclic antidepressants, Monoamine Oxidase inhibitors), orthopedic antipsychotic drugs, etc.
12. Subjects with previous administration of all clinical trial vaccines for Alzheimer's disease
13. Subjects who consented to lumbar puncture (LP) for Cerebrospinal Fluid (CSF) examination only check the following exclusion criteria

    - Subjects who are not contraindicated (e.g. platelet count <100,000/μL, lumbar deformity, etc.) for performing lumbar puncture. Subjects can participate in clinical trials even if they are contraindicated in performing a lumbar puncture.
14. Female subjects with childbearing potential who do not agree to contraception using a medically accepted method (complete celibacy; hormonal contraceptives: Levonorgestrel, Intrauterine system of Mirena, and Medroxyprogesterone; and surgical sterilizations: vasectomy, double tubectomy, double tubal ligation) during the clinical trial period and until 90 days after clinical trial end (stop).
15. Pregnant or lactating women
16. Subjects who participated in another clinical trial within 4 weeks before participation in this clinical trial
17. Subjects in less than 12 months after the administration of the Investigational product for this clinical trial
18. Subjects who participated in any clinical trial for Alzheimer type dementia treatment within 6 months at screening
19. Subjects who are judged by the investigator to be ineligible for participation in this clinical trial

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in SIB(Severe Impairment Battery) score after GV1001 administration for 24 weeks | Baseline, Week 26
  SIB includes 51 questions to assess cognition in an individual. SIB consists of nine symptom domains such as attention, language, orientation, memory, praxis, visuospatial perception, construction, social skills and orientating head to name. The possible total scores range from 0 to 100 with a higher score indicating greater cognitive function.
CIBIC-plus (Clinician Interview-Based Impression of Change-Plus) score after GV1001 administration for 24 weeks | Baseline, Week 26
  CIBIC-plus consists of 4 items: "Overall," "Mental and Cognitive Function," "Behavior," and "Daily Function." CIBIS, a 7-point severity assessment, is administered at baseline. CIBIC-plus is implemented at follow-up visits to evaluate the degree of change in overall functional status in 7 levels by referring to the CIBIS results evaluated at baseline. The overall clinical condition of the dementia patient is assessed based on information obtained from semi-structured interviews of patients and caregivers. The rater is independent, has clinical experience, and will evaluate the subjects after completing the training required for this study.

SECONDARY OUTCOMES:
Change from baseline in SIB(Severe Impairment Battery) score | Baseline, Week 6, and Week 14
  SIB includes 51 questions to assess cognition in an individual. SIB consists of nine symptom domains such as attention, language, orientation, memory, praxis, visuospatial perception, construction, social skills and orientating head to name. The possible total scores range from 0 to 100 with a higher score indicating greater cognitive function.
CIBIC-plus (Clinician Interview-Based Impression of Change-Plus) score after GV1001 administration | Baseline, Week 6, and Week 14
  CIBIC-plus consists of 4 items: "Overall," "Mental and Cognitive Function," "Behavior," and "Daily Function." CIBIS, a 7-point severity assessment, is administered at baseline. And CIBIC-plus is implemented at follow-up visits to evaluate the degree of change in overall functional status in 7 levels by referring to the CIBIS results evaluated at baseline. The overall clinical condition of the dementia patient is assessed based on information obtained from semi-structured interviews of patients and caregivers. The rater is independent, has clinical experience, and will evaluate the subjects after completing the training required for this study.
Change from baseline in K-MMSE(Korea Mini-Mental State Examination) score after GV1001 administration | Baseline, Week 6 week, Week 14, and Week 26
  K-MMSE assesses an individual's cognitive function by asking questions about time orientation, spatial orientation, memory registration, attention and calculation, memory recall, language, and space-time configuration. It creates the possible total score from 0 to 30, with a lower total score indicating greater severity in cognitive impairment.
Change from baseline in NPI-Q(Neuropsychiatric Inventory Questionnaire) score after GV1001 administration | Baseline, Week 6 week, Week 14, and Week 26
  NPI-Q consists of questions to evaluate degrees of behavioral disturbance in 12 domains. It includes delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, and appetite/eating. The severity scale has scores ranging from 1 to 3 points (1=mild and 3=severe) and the scale for assessing caregiver distress has scores ranging from 0 to 5 points (0=no distress and 5=extreme distress). The higher sum of the NPI-Q severity score represents greater severity of the individual's symptoms, and the higher sum of the NPI-Q distress score indicates greater severity of caregiver's distress associated with the symptoms.
Change from baseline in GDS(Global Deterioration Scale) score after GV1001 administration | Baseline, Week 6 week, Week 14, and Week 26
  GDS provides the stages for the severity of cognitive function of the individual with AD. It is brown down into seven stages (stage1=no cognitive decline and 7=very severe cognitive decline).
Change from baseline in ADCS-ADL-severe(Alzheimer's Disease Cooperative Study-Activities of Daily Living scale-severe) score after GV1001 administration | Baseline, Week 6 week, Week 14, and Week 26
  ADCS-ADL-severe consists of 19 items that can access the competence of individuals with AD in activities of daily living. The maximum possible total score is 54, with a higher score indicating lesser severity in AD.
Change from baseline in CDR-SOB(Clinical Dementia Rating Scale Sum of Boxes) score after GV1001 administration | Baseline, Week 6 week, Week 14, and Week 26
  CDR-SOB evaluates cognitive and functional performance in six domains related to AD including memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated from 0 to 5 points (0, 0.5, 1, 2, 3, 4, and 5) with a lower total score indicating severely impaired cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Kyounghee Seo, Study Director — Samsung Pharmaceutical Co., Ltd.

IPD SHARING:
Plan to Share IPD: No